CLINICAL TRIAL: NCT03815565
Title: Comparison Between Continuous Femoral Block With Levobupivacaine 0.125% and Ropivacaine 0.2% for Preoperative Analgesia, in Patients Over 70 Years Old, With Proximal Femoral Fractures: a Randomized, Double-blind Study
Brief Title: Continuous Femoral Block With Levobupivacaine 0.125% or Ropivacaine 0.2% in Elderly Patients With Femoral Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Municipal Miguel Couto (Other)
Responsible Party: Principal Investigator, Rafael Mercante Linhares, Head of Anesthesiology and Pain Medicine Department, Hospital Municipal Miguel Couto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 65821217.5.0000.8066
Record Dates: First submitted 2019-01-08; First posted 2019-01-24 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Femur Fracture; Hip Fractures
Keywords: analgesia; continuous; femoral block
MeSH Terms: conditions — Femoral Fractures; Hip Fractures; Agnosia

STUDY DESIGN:
Intervention Model Description: randomized
Who Masked: Participant, Investigator
Masking Description: Only the pharmacist chief knows which participant belongs to each arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- levobupivacaine 0.125% (Experimental): continuous femoral block with levobupivacaine 0.125%. Use of PCA pump with the following parameters: 5 ml/h; bolus 5 ml; lockout 30 minutes
  Interventions: Procedure: continuous femoral block
- ropivacaine 0.2% (Active Comparator): continuous femoral block with ropivacaine 0.2%. Use of PCA pump with the following parameters: 5 ml/h; bolus 5 ml; lockout 30 minutes
  Interventions: Procedure: continuous femoral block

INTERVENTIONS:
Procedure: continuous femoral block — infusion of anesthetic by PCA pump

SUMMARY:
This study evaluates the continuous femoral block between levobupivacaine 0.125% and ropivacaine 0.2% in patients with proximal femoral fracture.These patients will be divided into 2 groups of 35 patients, one L group (levobupivacaine 0.125%) and one R group (ropivacaine 0.2%) distributed randomly, receiving continuous infusion through patient controlled analgesia (PCA) pump with the following parameters: infusion 5 ml / h, bolus 5 ml, lockout 30 min.

DETAILED DESCRIPTION:
Pain is associated with neurohormonal stress, myocardial ischemia and delayed mobilization, thus being able to increase the hospitalization time and associated with increased postoperative mortality. Regional anesthesia through simple or continuous femoral nerve block are options for analgesia in patients with femoral fracture, as well as analgesia by venous opioids. A potential benefit of regional anesthesia is precisely to avoid the use of opioids and other general anesthetics, which in turn are also closely related to postoperative delirium. Continuous femoral block, since the preoperative period, is associated with the reduction of acute pain and opioid consumption, in patients with femoral neck fractures. There are few studies available in the literature comparing analgesic equipotency between levobupivacaine and ropivacaine in peripheral nerve blocks. In none of them, the peripheral analgesia in the femoral nerve, for proximal femoral fracture was compared.

ELIGIBILITY:
Inclusion Criteria:

* 70 years old or more
* patients with femur fracture
* physical status risk American Society of Anesthesiologists (ASA) P1 - P3

Exclusion Criteria:

* physical status ASA P4
* patients with BMI > 35
* systemic infection
* Injury or infection at the site of installation of the femoral perineural catheter
* Catheter displacement of the perineural site
* Montreal Cognitive Assessment (MoCA) < 26
* Patients operated before 24 hours of hospital admission

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2020-08-08 (Estimated); Study Completion 2021-01-08 (Estimated)

PRIMARY OUTCOMES:
intensity of individual pain episodes | 6 hours after hospital admission
  Self report pain intensity in the preoperative period. Scored 0-10 (0 = no pain; 10 = pain as bad as can be)

SECONDARY OUTCOMES:
Number of PCA firing | 72 hours
  in each patient at time of evaluation of pain
Degree of satisfaction with analgesic therapy | up to 72 hours - at the moment of surgery; or at the end of 72 hours
  using the 5-point rating scale (very dissatisfied, dissatisfied, neutral, satisfied or very pleased)
Quality of sleep | up to 72 hours
  very good, good, bad and very bad
the cost of analgesic therapy | up to 72 hours
  including catheters, PCA and medication in each patient
adverse event | up to 72 hours
  paresthesia, nausea, vomiting, ringing in the ear, metallic taste, convulsion or cardiac arrest

CONTACTS AND LOCATIONS:
Locations (1):
- Rafael M Linhares, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
after the finish of the study

REFERENCES:
- [Background] Joshi G, Gandhi K, Shah N, Gadsden J, Corman SL. Peripheral nerve blocks in the management of postoperative pain: challenges and opportunities. J Clin Anesth. 2016 Dec;35:524-529. doi: 10.1016/j.jclinane.2016.08.041. Epub 2016 Oct 20. PMID 27871587
- [Result] Ritcey B, Pageau P, Woo MY, Perry JJ. Regional Nerve Blocks For Hip and Femoral Neck Fractures in the Emergency Department: A Systematic Review. CJEM. 2016 Jan;18(1):37-47. doi: 10.1017/cem.2015.75. Epub 2015 Sep 2. PMID 26330019
- [Result] Morrison SR, Magaziner J, McLaughlin MA, Orosz G, Silberzweig SB, Koval KJ, Siu AL. The impact of post-operative pain on outcomes following hip fracture. Pain. 2003 Jun;103(3):303-311. doi: 10.1016/S0304-3959(02)00458-X. PMID 12791436
- [Result] Szucs S, Iohom G, O'Donnell B, Sajgalik P, Ahmad I, Salah N, Shorten G. Analgesic efficacy of continuous femoral nerve block commenced prior to operative fixation of fractured neck of femur. Perioper Med (Lond). 2012 Jun 27;1:4. doi: 10.1186/2047-0525-1-4. eCollection 2012. PMID 24764520